CLINICAL TRIAL: NCT03269084
Title: Type 1 Diabetes Prediction and Prevention (DIPP) Study
Acronym: DIPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riitta Veijola (Other)
Collaborators: Oulu University Hospital (Other); University of Turku (Other); Turku University Hospital (Other Government); Tampere University (Other); Tampere University Hospital (Other); Juvenile Diabetes Research Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor-Investigator, Riitta Veijola, Professor of Pediatrics, University of Oulu
Organization: University of Oulu (Other)
Other Study IDs: 1-SRA-2016-342-M-R
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children at HLA-conferred risk for T1D
  Interventions: Other: No intervention. DIPP is an observational study.

INTERVENTIONS:
Other: No intervention. DIPP is an observational study.

SUMMARY:
The Type 1 Diabetes Prediction and Prevention (DIPP) Study in Finland is a population-based long-term clinical follow-up study established since 1994 in three university hospitals in Finland to understand the pathogenesis of type 1 diabetes (T1D), predict the disease, and find preventive treatment.

DETAILED DESCRIPTION:
Briefly, cord blood samples are collected and HLA-DR-DQ genotypes are determined from newborn babies. Families with a newborn baby carrying a DR-DQ genotype associated with increased risk for T1D are invited to participate in regular follow-up at the age of 3, 6, 9, 12, 18 and 24 months, and thereafter once a year until the age of 15 years or until T1D is diagnosed. Clinical details including maternal diet during pregnancy and lactation and child's diet starting from the age of 3 months are recorded, blood samples are collected, and serum autoantibodies associated with development of T1D are measured. Children who develop beta-cell specific autoimmunity are followed more intensively with measurements of glucose metabolism parameters such as glycated haemoglobin A1c (HbA1c), oral glucose tolerance tests (OGTT) and intravenous glucose tolerance tests (IVGTT). In the DIPP Study more than 1000 children have developed multiple islet autoantibodies and more than 450 of these have progressed to clinical T1D. It has been estimated that 5% of children in the follow-up will develop T1D and 60% of future T1D cases will be reached by the current screening and follow-up strategy.

ELIGIBILITY:
Inclusion Criteria:

* Newborn babies with HLA-conferred genetic susceptibility to type 1 diabetes born in three University Hospitals in Finland

Exclusion Criteria:

* Newborn babies without HLA-conferred genetic susceptibility to type 1 diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Since November 1994 the Finnish Type 1 Diabetes Prediction and Prevention (DIPP) Study has screened 206,707 newborns for HLA-conferred genetic susceptibility for T1D (Figure 1., data as of March 2015). A total of 16,193 children have started clinical follow-up with regular study visits and systematic collection of longitudinal blood and stool samples. Altogether more than 1000 children have seroconverted to positivity for multiple islet autoantibodies (ICA included). A total of 461 children and adolescents have progressed to clinical T1D with DIPP follow-up from birth until diagnosis. Currently there are 7158 children between 3 months and 15 years of age taking part in the DIPP Study follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Estimated)
Dates: Start 1994-11-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Positivity for at least one islet autoantibody | December 31, 2021
  ICA, IAA, GADA, IA-2A or ZnT8A
Clinical diagnosis of type 1 diabetes | December 31, 2021
  Hyperglycemia as defined by WHO

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Veijola, MD PhD, Principal Investigator — University of Oulu, Oulu University Hospital; Mikael Knip, MD PhD, Principal Investigator — University of Helsinki, Tampere University Hospital; Jorma Toppari, MD PhD, Principal Investigator — University of Turku, Turku University Hospital; Kalle Kurppa, MD PhD, Principal Investigator — Tampere University; Heikki Hyöty, MD PhD, Principal Investigator — Tampere University; Johanna Lempainen, MD PhD, Principal Investigator — University of Turku
Locations (3):
- Finland (3):
  - University of Oulu and Oulu University Hospital, Oulu
  - University of Tampere and Tampere University Hospital, Tampere
  - University of Turku and Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kyronniemi A, Valtanen T, Koskenniemi J, Vahasalo P, Harkonen T, Ilonen J, Toppari J, Knip M, Veijola R. Extremely Early Appearance of Islet Autoantibodies in Genetically Susceptible Children. Pediatr Diabetes. 2023 Dec 11;2023:9973135. doi: 10.1155/2023/9973135. eCollection 2023. PMID 40303239